CLINICAL TRIAL: NCT04267601
Title: A Non-interventional, Single Group, Open-label, Multicenter Observational Study to Evaluate the Efficacy and Safety of Anagliptin in Type 2 Diabetic Patients With Other DPP4is as Mono or Combination Therapy With Insufficient Glucose Control
Brief Title: Korean Observational Study to Evaluate the Efficacy and Safety of Anagliptin Switching From Other DPP4is in type2 DM
Acronym: SSUG
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: JWP-GDL-402
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — anagliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anagliptin — Anagliptin treatment for 24weeks

SUMMARY:
This study was designed as a non-interventional, single-group, open-label, multicenter observational study for patients with type 2 diabetes in the real world clinical setting.

DETAILED DESCRIPTION:
Subjects will visit the site on the 12th week (Visit 2) and 24th week (Visit 3) from the registration date (Visit 1) to confirm the efficacy and safety.

Primary endpoint

- HbA1c change after 24 weeks treatment

Secondary endpoint

* Average rate of change in HbA1c after baseline
* Ratio of subjects with HbA1c<7% after 24 weeks
* Ratio of subjects with HbA1c<6.5% after 24 weeks
* Subgroup analysis by gender, age, BMI, medical history, renal function, liver function, conventional DPP4 inhibitors therapy, concomitant Oral Antidiabetic Drug, duration of disease

Safety endpoint : Adverse Event

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age at the time of consenting
* Understands and is willing to sign an informed consent form (ICF)
* HbA1c≥7.0%
* within 7days before registration, continuing other DPP4is alone or combined therapy for than 8 weeks

Exclusion Criteria:

* Prior exposure to Anagliptin

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic patients with other DPP4is as mono or combination therapy with insufficient glucose control
Sampling Method: Non-Probability Sample
Enrollment: 2448 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of HbA1C | after 24weeks treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Bucheon ST. Mary's hopsital, Bucheon-si, South Korea

IPD SHARING:
Plan to Share IPD: No